CLINICAL TRIAL: NCT05614141
Title: Investigation of the Effects of Virtual Reality Exercises Combined With Robot-assisted Walking Training on Individuals With Subacute Stroke on Cognitive Functions, Activities of Daily Living and Quality of Life.
Brief Title: Investigation of the Effects of Robot Assisted Gait Training With Virtual Reality on Cognitive Functions in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Murat Akıncı, MSc PT, Ankara Yildirim Beyazıt University
Other Study IDs: Lokomat Cognitive
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Exoskeleton Device; Locomotion; Stroke
Keywords: Lokomat; Augmented Performance Feedback
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group
  Interventions: Device: Lokomat Augmented Performance Feedback; Other: Conventional Physiotherapy
- Control Group
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Device: Lokomat Augmented Performance Feedback — All participants will exercise with Lokomat Augmented Performance Feedback for six weeks. Augmented Performance Feedback has different virtual reality games.
  Groups: Study Group
Other: Conventional Physiotherapy — Conventional physiotherapy includes stretching, strengthening, balance, coordination and walking exercises under the guidance of a physiotherapist.

SUMMARY:
It was planned to examine the effects of robot-assisted walking training supported by virtual reality on cognitive functions, quality of life and activities of daily living in individuals with subacute stroke. In this context, only conventional physiotherapy was applied to one group, while the other group was given exercises with Lokomat in addition to conventional physiotherapy.

DETAILED DESCRIPTION:
According to the definition of the World Health Organization, stroke is a clinical syndrome characterized by the rapid establishment of signs and symptoms of focal loss of cerebral function for no apparent reason other than vascular causes. Symptoms last longer than twenty-four hours or may result in death. Stroke is the second leading cause of death in the world and the first cause of disability and loss of work force. Many stroke survivors are dependent on someone else for some part of their daily lives, have limitations in their daily and social activities, and have significantly lost their quality of life. Cognitive disorders after stroke are manifested by difficulties in information processing due to brain damage. The most common cognitive effects in stroke; attention, memory, orientation, executive dysfunction and aphasia.

For cognitive rehabilitation it is known that Lokomat combined virtual reality applications is more effective than Lokomat exercises without virtual reality in individuals with chronic stroke. Our research aims to contribute to the literature by revealing the cognitive functions, ADL and quality of life of locomotive exercises together with virtual reality in individuals with subacute stroke.

Our research will be carried out in the Robotic Rehabilitation Laboratory of Physical Therapy and Rehabilitation Hospital in Ankara City Hospital. The population of the study is the stroke clinics of the same hospital. Individuals with subacute stroke who volunteered to participate in the study will be included in the study. All patients will receive conventional physiotherapy five days a week for six weeks, and the study group will receive with Lokomat three times a week in addition to conventional physiotherapy. The patients will be evaluated by a therapist other than the practitioner before and after the treatment in two groups, one of which is the study group and the other is the control group.

ELIGIBILITY:
Inclusion Criteria:

* First Stroke
* Subacut stroke (from 21 days to 180 days)
* Can do Lokomat exercises

Exclusion Criteria:

* incompatibility to lokomat (Femur lenght problems, severe cognitive impairment, excess weight etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research will be carried out with individuals with subacute stroke. Participation in the research is based on a voluntary basis.
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
MOCA Score | 6 weeks after treatment
  Montreal Cognitive Assessment (MOCA) assesses eight cognitive functions. These are attention and concentration, executive functions, memory, language, visual structuring, abstract thinking, computation, and orientation.

SECONDARY OUTCOMES:
Lawton&Brody Score | 6 weeks after treatment
  Instrumental Activities of Daily Living (Lawton&Brody Score) consists of 8 questions covering activities such as using the phone, shopping, using public transport, doing daily housework, preparing meals, and traveling. If the patient score is between 0-8 points, fully dependent, between 9-16 points semi-dependent, between 17-24 points is considered fully independent.
SS-QOL Score | 6 weeks after treatment
  The Stroke-Specific Quality of Life Scale is specially designed for stroke patients. It consists of 49 items covering 12 domains that measure quality of life. It measures in many fields such as upper extremity functions, visual functions, speech, domestic roles, social roles, mobility, psychological state, work productivity, self-care, perception, memory, and personality. High scores indicate better quality of life. The maximum score is 245.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided